CLINICAL TRIAL: NCT02278575
Title: Clinical Effect of Atenativ Treatment on Uterine Blood Flow and the Amount of Atenativ Needed to Maintain a Normal Antithrombin Lvels During Two Weeks in Early and Severe Preeclampsia
Brief Title: Atenativ Effect on Uterine Blood Flow and Preeclampsia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: impossible to recruit participants due to organization changes
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Octapharma (Industry)
Responsible Party: Principal Investigator, Margareta Hellgren, professor, MD, PhD, Vastra Gotaland Region
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EudraCT 2012-005770-57
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Antithrombin III Deficiency
Keywords: antithrombin, Atenativ, preeclampsia, blood flow.
MeSH Terms: conditions — Antithrombin III Deficiency; Pre-Eclampsia | interventions — Antithrombin III

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Consisting of treatment with Atenativ (Other): During two weeks antithrombin concentrate(Atenativ) will be administered in order to maintain normal levels of antithrombin
  Interventions: Drug: Atenativ

INTERVENTIONS:
Drug: Atenativ — intravenous transfusion
  Other Names: antithrombin concentrate

SUMMARY:
The study will be an open controlled pilot study of 6 patients with early-onset severe preeclampsia. Patients will receive Atenativ in addition to conventional therapy The patients will be followed up within the study until three days after delivery. Laboratory analyses and uterine and umbiliacal blood flow will be determined.

DETAILED DESCRIPTION:
The study will be an open controlled pilot study of 6 patients with early-onset severe preeclampsia. Patients will receive Atenativ in addition to conventional therapy The patients will be followed up within the study until three days after delivery. In addition to conventional therapy, i.v. administration of Atenativ will be given in a dosage aimed to raise the plasma level of AT initially to 120% (1.2 kIU/L) The goal is to achieve and maintain plasma activity of about 100% during two weeks. The dose of Atenativ is based on the actual plasma level of AT measured 2 hours before the dose. During the first two days of treatment plasma samples will be drawn for the measurement of AT activity twice a day, once before and 12 hours after infusion in order to monitor the dosage. Thereafter and until study discontinuation AT will be measured once a day. The treatment will continue for two weeks if plasma AT III is below 100% (1.0 kIU/L).Uterine blood flow is measured before, during and after the AT infusion. Demographic data, medical history and other background data (age, weight, height, gestational week, smoker or not, gravidity, parity, previous hypertension, previous medication etc) will be recorded in order to ensure that the inclusion criteria are met and to verify patient identity and inclusion status. The week of gestation when the patient is included in the study as well as the week of gestation at delivery is recorded.

The type of delivery (vaginal or caesarean section as well as planned or acute) will also be recorded.. General haemostatic parameters are to be analyzed before start of treatment and then every day during treatment and thereafter at least twice a week. Special haemostatic parameters are Placental growth factor, S-Flt-1, VEGF and Syndecan-1. They will be sampled before start of treatment and during treatment once a week. The samples will be collected and frozen and not analyzed before the termination of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant woman in gestational week 23+0 - 29+0
2. Severe preeclampsia as defined by international criteria (1,2)

   * Blood pressure >160/110 mmHg (measured twice 30 minutes apart). proteinuria (>5 .0 g/L per 24 hours or >3 + labstick in at least two random samples six hours apart) after 20th gestational week.
   * Blood pressure >140/90 mmHg and proteinuria >5.0 g/24 h.
   * preeclampsia ( blood pressure > 140/90 and proteinuria >0.3 g/24 h) with IUGR or subjective symptoms as epigastic pain (HELLP), headache, dizziness or visual disturbancies, oligouri < 600 ml/24 h, coagulation disturbancies.
3. AT level <0.8 kIE/L

   -

Exclusion Criteria:1. History of congenital AT deficiency 2. Severe preeclampsia with demand on acute delivery within 24 hours according to the investigators judgments 3. Concomitant administration of anticoagulants and platelet inhibitors within 2 weeks 4. Chronic renal disease 5. Diabetes melittus or gestational diabetes 6. Intrauterine fetal death 7. Participation in another clinical study 8. Multiple pregnancies

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Blood flow in uterin and umbilical artery | up to day 14

SECONDARY OUTCOMES:
fetal outcome | at birth
  CTG, blood flow, Apgar score, birthweight
bleeding complications | during pregnancy and at delivery
  measurements of bleeding before and after placenta delivery

OTHER OUTCOMES:
Biomarkers of endothelial damage | up to day 14
  S-Flt-1, VEGF,Syndecan-1
Atenativ concentrate | treatment during 2 weeks
  amount needed to maintain normal antithrombin levels

CONTACTS AND LOCATIONS:
Overall Officials: Margareta Hellgren, MD,PhD,prof, Principal Investigator — department Obstetrics, Sahlgrenska University Hospital
Locations (1):
- Dept Obstetrics, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
extern monitoring by Gothia Forum

REFERENCES:
- [Result] Heilmann L, Rath W, Pollow K. Hemostatic abnormalities in patients with severe preeclampsia. Clin Appl Thromb Hemost. 2007 Jul;13(3):285-91. doi: 10.1177/1076029607299986. PMID 17636190
- [Result] Weenink GH, Treffers PE, Vijn P, Smorenberg-Schoorl ME, ten Cate JW. Plasma antithrombin III levels in pre-eclampsia. Clin Exp Hypertens B. 1983;2(1):145-62. doi: 10.3109/10641958309023467. PMID 6872275
- [Result] Aghai E, Brunstein J, Quitt M, Abramovici H, Froom P. Antithrombin III levels in preeclampsia. Isr J Med Sci. 1990 Mar;26(3):142-3. PMID 2329037
- [Result] Hellgren M, Hagnevik K, Robbe H, Bjork O, Blomback M, Eklund J. Severe acquired antithrombin III deficiency in relation to hepatic and renal insufficiency and intrauterine fetal death in late pregnancy. Gynecol Obstet Invest. 1983;16(2):107-18. doi: 10.1159/000299230. PMID 6618278
- [Result] Hellgren M, Javelin L, Hagnevik K, Blomback M. Antithrombin III concentrate as adjuvant in DIC treatment. A pilot study in 9 severely ill patients. Thromb Res. 1984 Aug 15;35(4):459-66. doi: 10.1016/0049-3848(84)90237-8. No abstract available. PMID 6484893
- [Result] Maki M, Kobayashi T, Terao T, Ikenoue T, Satoh K, Nakabayashi M, Sagara Y, Kajiwara Y, Urata M. Antithrombin therapy for severe preeclampsia: results of a double-blind, randomized, placebo-controlled trial. BI51.017 Study Group. Thromb Haemost. 2000 Oct;84(4):583-90. PMID 11057854
- [Result] Kobayashi T, Terao T, Ikenoue T, Sameshima H, Nakabayashi M, Kajiwara Y, Maki M; BI 51 017 Study Group. Treatment of severe preeclampsia with antithrombin concentrate: results of a prospective feasibility study. Semin Thromb Hemost. 2003 Dec;29(6):645-52. doi: 10.1055/s-2004-815632. PMID 14719181
- [Result] Paternoster DM, Fantinato S, Manganelli F, Nicolini U, Milani M, Girolami A. Recent progress in the therapeutic management of pre-eclampsia. Expert Opin Pharmacother. 2004 Nov;5(11):2233-9. doi: 10.1517/14656566.5.11.2233. PMID 15500369
- [Result] Sameshima H, Kodama Y, Ikenoue T, Kajiwara Y. Antithrombin improves fetal condition in women with severe pre-eclampsia before 32 weeks of gestation; a randomized, double-blind, placebo-controlled trial. J Obstet Gynaecol Res. 2008 Feb;34(1):34-9. doi: 10.1111/j.1447-0756.2007.00677.x. PMID 18226126